CLINICAL TRIAL: NCT02370264
Title: Screening for Musculoskeletal Impairments and Quality of Life in Individuals Post-Treatment for Breast Cancer
Brief Title: Questionnaires in Identifying Upper Extremity Function and Quality of Life After Treatment in Patients With Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not progressing toward scientific goals
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1B-12-4; NCI-2014-01849 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HS-12-00578-CR002; HS-12-00578; 1B-12-4 (Other: USC Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2015-02-17; First posted 2015-02-24 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Musculoskeletal Complication; Recurrent Breast Carcinoma; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer; Therapy-Related Toxicity
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (musculoskeletal screening, quality of life) (Experimental): Patients complete the DASH and FACT-B questionnaires over 30-45 minutes.
  Interventions: Procedure: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Medical Chart Review

INTERVENTIONS:
Procedure: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Medical Chart Review — Ancillary studies
  Other Names: Chart Review

SUMMARY:
This pilot clinical trial studies questionnaires in identifying arms, shoulder, and neck (upper extremity) function and quality of life after treatment in patients with breast cancer. Patients may experience arms, shoulder, and neck impairments that negatively affect their functioning and quality of life after cancer-related treatment. Studying upper extremity function and quality of life in patients after breast cancer treatment may help doctors determine the prevalence and severity of long-term functional impairments and the relationship between the perception of impairments due to breast cancer treatment and its' impact on quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To characterize patients' upper extremity functionality (using the Disabilities of the Arm, Shoulder and Hand [DASH] questionnaire) and their perception of quality of life (using the Functional Assessment of Cancer Therapy-Breast [FACT-B] questionnaire) one to ten years after breast cancer surgery and compare it to the general population.

II. To investigate whether patients' upper extremity functionality and their perception of quality of life after completion of breast cancer treatment changes over the duration of time between 1 -10 years after breast cancer surgery.

III. To characterize patient perception of the impact of breast cancer on their quality of life in relation to current upper-extremity functionality 1-10 years after breast cancer surgery.

IV. To characterize patients' upper extremity functionality (using the DASH questionnaire) and their perception of the impact of breast cancer on their quality of life (using the FACT-B questionnaire) in a sub group of individuals with stable metastatic breast cancer 1-10 years after initial diagnosis and surgery.

SECONDARY OBJECTIVES:

I. To assist the multidisciplinary team to identify musculoskeletal barriers (if any) that impact a patient's long-term recovery with respect to the breast cancer treatments they have received.

II. To assist in developing and implementing a physical therapy component within the Personalized Medicine to Breast Cancer Care Plan; this includes early detection of potential physical barriers, physical therapy intervention models, and development of survivorship planning for cancer-related musculoskeletal impairments.

OUTLINE:

Patients complete the DASH and FACT-B questionnaires over 30-45 minutes.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a history of breast cancer surgery either lumpectomy, mastectomy, axillary node dissection or sentinel node biopsy at least one year ago and received either radiation therapy or chemotherapy or both
* Patients with no active disease; (as defined as no detectable disease)
* Patients with stable metastatic disease which is defined as (metastatic tumor demonstrates no increase in volume, tumor size or diameter and no evidence of new lesions, have been identified during last assessment by medical oncologist/radiologist or surgeons)
* Signed informed consent

Exclusion Criteria:

* Survivors of breast cancer that have not received either breast surgery or radiation therapy
* Patients with known cognitive impairments
* Individuals with progressive metastatic disease in which the tumor has increased in size, volume and diameter or evidence of new lesions, as noted by medical oncologists, radiologists and surgeons
* individuals who are non-ambulatory
* Women who self-report to be pregnant

  * As this is an observational study, we will not be performing a pregnancy test, participants will be asked if they are or are not pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2015-09-02 (Actual); Study Completion 2016-10-21 (Actual)

PRIMARY OUTCOMES:
Patients' upper extremity functionally 1 to 10 years after treatment using DASH score | Baseline
  DASH scores ranges from 0-100 with 1 being the least disability and 100 indicating the most disability. Means and standard deviation of the DASH will be calculated separately for patients with stable metastatic disease and those without metastatic diseases. These means will be compared with the general population.
Patients' perception of quality of life (QOL) 1 to 10 years after treatment using the FACT-B score | Baseline
  The total FACT-B score ranks from 0-144, with a high score indicating a better QOL. Means and standard deviation of the FACT-B will be calculated separately for patients with stable metastatic disease and those without metastatic diseases. These means will be compared with the general population.
Discrepancy between the presence of physical impairments and patients' perception of QOL assessed using DASH and FACT-B scores | Baseline
  Using the distribution of the DASH and FACT-B scores reported in general population based studies, the percentile rank of each patient's DASH or FACT-B score will be calculated. Given that a higher DASH score indicates worse disability while a higher FACT-B score means a better quality of life, the percentile ranks for DASH will be subtracted from 100 and the remainder will be used as the percentile ranks for DASH for analyses purposes.
Time effect in the DASH score 1 to 10 years following treatment | Baseline
  A linear regression model will be used to examine whether there is a time effect in the DASH score with DASH being the independent variable and time after treatment being the predictive variable. Other factors that will also be investigated as affecting DASH score will include whether or not a patient had full axillary lymph node dissection or sentinel lymph node dissection, or whether or not a patient received radiation therapy or chemotherapy, etc. Interaction between these main effects and time will be included to assess differences in time effect.
Time effect in the FACT-B score 1 to 10 years following treatment | Baseline
  A linear regression model will be used to examine whether there is a time effect in the FACT-B score with FACT-B score being the independent variable and time after treatment being the predictive variable. Other factors that will also be investigated as affecting FACT-B score will include whether or not a patient had full axillary lymph node dissection or sentinel lymph node dissection, or whether or not a patient received radiation therapy or chemotherapy, etc. Interaction between these main effects and time will be included to assess differences in time effect.

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Perdomo, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States